CLINICAL TRIAL: NCT05034627
Title: A Phase I, Open-Label, Dose Finding Study of Calaspargase Pegol-Mnkl in Combination With Cobimetinib in Locally-Advanced or Metastatic Pancreatic Cancer
Brief Title: Calaspargase Pegol-Mnkl and Cobimetinib for the Treatment of Locally Advanced or Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Genentech, Inc. (Industry); Servier Pharmaceuticals, LLC (Unknown)
Responsible Party: Principal Investigator, Charles D Lopez, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00022141; NCI-2021-09061 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00022141 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma; Metastatic Pancreatic Adenocarcinoma; Stage II Pancreatic Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8; Stage IIB Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy; calaspargase pegol; Asparaginase; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (calaspargase pegol-mknl, cobimetinib) (Experimental): Patients receive calaspargase pegol-mknl IV over 1 hour on day 1 and cobimetinib PO QD on days 1-14. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may also undergo a biopsy 14 days prior to starting therapybefore cycle 1, day 1 and again on day 14 of cycle 2, day 15 per the investigator's discretion, with an additional optional biopsy at the time of disease progression.
  Interventions: Procedure: Biopsy; Drug: Calaspargase Pegol-mknl; Drug: Cobimetinib

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Drug: Calaspargase Pegol-mknl — Given IV
  Other Names: Asparaginase (Escherichia coli Isoenzyme II), Conjugate with alpha-(((2,5-Dioxo-1-pyrrolidinyl)oxy)carbonyl)-omega-methoxypoly(oxy-1,2-ethanediyl); Asparlas; Calaspargase Pegol; EZN-2285; SC-PEG E. Coli L-Asparaginase; Succinimidyl Carbonate Monomethoxypolyethylene Glycol E. coli L-Asparaginase
Drug: Cobimetinib — Given PO
  Other Names: Cotellic; GDC-0973; MEK Inhibitor GDC-0973; XL518

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of calaspargase pegol-mknl in combination with cobimetinib in treating patients with pancreatic cancer that has spread to nearby tissue or lymph nodes (locally advanced) or has spread to other places in the body (metastatic). Cobimetinib attacks a protein called MEK that has been known to stimulate cells that promote the growth of cancer cells in the body. Calaspargase pegol-mknl is an enzyme that converts the amino acid L-asparagine into aspartic acid and ammonia. Many types of cancer cell rely on the amino acid L-asparagine, and depleting this amino acid with calaspargase pegol-mknl starves cancer cells of this nutrient. Attacking the MEK protein with cobimetinib is thought to further prevent cancer cells from using this amino acid, causing them to die. Giving calaspargase pegol-mknl in combination with cobimetinib may help control the disease in patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) of calaspargase pegol-mknl in combination with cobimetinib.

SECONDARY OBJECTIVES:

I. To assess the safety of calaspargase pegol-mknl in combination with cobimetinib.

II. To assess preliminary response to treatment with calaspargase pegol-mknl and cobimetinib.

III. To monitor levels of plasma asparaginase.

EXPLORATORY OBJECTIVE:

I. To evaluate therapy induced changes in the tumor and tumor ecosystem.

OUTLINE: This is a dose-escalation study.

Patients receive calaspargase pegol-mknl intravenously (IV) over 1 hour on day 1 and cobimetinib orally (PO) once daily (QD) on days 1-14. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may also undergo a biopsy before cycle 1, day1 and again on cycle 2 day 15 per the investiagator's discretion, with an additional biopsy at the time of disease progression.

After completion of study intervention, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant must provide written informed consent before any study-specific procedures or interventions are performed
* Participants are >= 18 years old at the time of informed consent. Both men and women of all races and ethnic groups will be included
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Histologically or cytologically-proven adenocarcinoma of the exocrine pancreas with locally advanced or metastatic disease
* Must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* Must have at least one disease lesion that is amenable to biopsy procedures performed per institutional standards
* Must have progressed on, been intolerant to, or refused systemic therapy that is consistent with institutional standards (e.g., Gemcitabine-based, or fluorouracil, irinotecan, leucovorin and oxaliplatin [FOLFORINOX])
* Must not have received any systemic therapy or other investigational agents within 30 days or 5 half-lives (whichever is longer) from first dose of study therapy

  * This requirement is waived for patients receiving cobimetinib or other investigational agent(s) as part of participation in NCT04005690, provided that all prior study-drug-related toxicities pertaining to NCT04005690 have resolved to grade =< 1 prior to initiating study intervention
* Hemoglobin: >= 8.5 g/dL with no blood transfusion within 14 days of starting treatment
* White blood cells (WBC): > 2.5 x 10^9/L
* Absolute neutrophil count (ANC): >= 1.2 x 10^9/L (> 1200 per mm^3)
* Platelet count: >= 90 x 10^9/L (> 90,000 per mm^3)
* Creatinine =< 1.5 x upper limit of normal (ULN), or measured or calculated creatinine clearance >= 60 mL/min/1.73 m^2 for participants with creatinine levels > 1 x institutional (ULN)
* Serum bilirubin: =< 1.5 x institutional ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT): =< 2.5 x ULN
* Participants must be able to take anticoagulant therapy while receiving calaspargase pegol-mknl
* Participants of childbearing potential (POCBP) must agree to abstain from sexual intercourse or use effective non-hormonal methods of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy (because calaspargase pegol can render hormonal contraceptives ineffective)
* POCBP may participate provided they have a negative serum pregnancy test at screening and a negative serum OR urine pregnancy test within 7 days of starting treatment

Exclusion Criteria:

* Concomitant use of other anti-cancer therapy (chemotherapy, immunotherapy, hormonal therapy (hormone replacement therapy is acceptable), radiotherapy (except for palliative), biological therapy or other novel agent) or live virus and live bacterial vaccines while receiving study medication
* Prior treatment with an L-asparaginase therapy
* Known severe hypersensitivity to calaspargase pegol-mknl (or equivalent) or to cobimetinib (or equivalent), or to any excipient of these medicinal products, or history of allergic reactions attributed to compounds of similar chemical or biologic composition to calaspargase pego-mknl or cobimetinib
* Use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir), known strong CYP3A inducers (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil) within 7 days of prior to initiating study treatment or on going requirement for these medications
* Uncontrolled serious thrombosis
* Uncontrolled severe or symptomatic coagulopathy; exclude if:

  * Prothrombin time (PT) >= 1.5 x ULN, or
  * International normalized ratio (INR) >= 1.5 x ULN, or
  * Fibrinogen =< 0.66 x LLN
* Known history of chronic pancreatitis or recurrent acute pancreatitis, or at time of screening evidence of acute pancreatitis, defined by at least two of the following:

  * Clinical symptoms of upper abdominal pain
  * Serum amylase or lipase that is >= 3 x ULN
  * Imaging evidence (computed tomography [CT], magnetic resonance imaging [MRI], ultrasonography)
* Significant cardiac disease within 6 months prior to start of study treatment, including any of the following:

  * New York Heart Association class III or IV,
  * Congestive heart failure, acute coronary syndrome, and/or stroke, or
  * Left ventricular ejection fraction (LVEF) < 40% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan obtained within 28 days prior to start of study treatment
* Known risk factors for ocular toxicity, consisting of any of the following:

  * History of serous retinopathy
  * History of retinal vein occlusion (RVO)
  * Evidence of ongoing serous retinopathy or RVO at screening
* Uncontrolled hypertension, or hypertension that cannot otherwise be clinically managed before initiating study therapy
* Participant is known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally
* Participant has active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
* Participant has corrected QT (QTc) interval (i.e., Fridericia's correction [QTcF]) >= 450 ms or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) at screening
* Psychiatric illness/social situations that would limit compliance with study requirements
* Any concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, etc.)
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 90 days after the last dose of trial treatment
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | Up to cycle 2 day 21 (1 cycle = 21 days)
  Defined as any treatment-related grade >= 3 non-hematological or hematological adverse events. The incidence of DLT at each dose level will be summarized using the proportion and exact binomial confidence interval. Dose-limiting toxicities will specifically be reported for the DLT evaluation period using the maximum tolerated dose (MTD)-evaluable population. The MTD will be identified using isotonic regression.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) and serious AEs | Up to 30 days after last dose of study intervention
  Evaluated by Common Terminology Criteria for Adverse Events version 5.0.
Objective response rate (ORR) | Up to 6 months after initiating study intervention
  Evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Overall response will be summarized descriptively. ORR will be estimated with 95% confidence interval. The confidence interval will be calculated based on the exact method for binomial distributions.
Disease control rate (DCR) | Up to 6 months after initiating study intervention
  Evaluated using RECIST version 1.1. An estimate of DCR will be measured and reported with 95% exact confidence interval. Participants who achieve a complete response, partial response, or stable disease for at least 6 months on the current protocol will be qualified as deriving benefit from therapy and will count towards the DCR measurement.
Mean plasma asparaginase activity | Up to 6 cycles from initiating study intervention (1 cycle = 21 days)
  Will be reported with 95% confidence interval.

OTHER OUTCOMES:
Therapy induced changes in the tumor and tumor ecosystem | Up to 6 cycles from completing study intervention (1 cycle = 21 days)
  Descriptive summary of cellular and molecular assays.

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Lopez, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States